CLINICAL TRIAL: NCT04875078
Title: UVA-1 for Treatment of Skin Tightening and Improvement of Hand Function in Scleroderma: a Randomized, Intra-patient, Dominant/non-dominant Hand Clinical Trial.
Brief Title: UVA-1 for Treatment of Skin Tightening and Improvement of Hand Function in Scleroderma
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Christopher B Hansen, Dr., University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB_00134454
Record Dates: First submitted 2021-04-30; First posted 2021-05-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Intervention Model Description: Treated hand compared to non-treated hand
Who Masked: Investigator
Masking Description: Investigator will be blinded to which hand was treated, and be the blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- UVA-1 Treated hand (Experimental): This hand will be treated with UVA-1 phototherapy.
  Interventions: Device: UVA-1 Phototherapy
- The untreated hand (No Intervention): This hand will be gloved when the patient undergoes UVA-1 phototherapy treatments.

INTERVENTIONS:
Device: UVA-1 Phototherapy — UVA-1 Phototherapy treatments
  Arms: UVA-1 Treated hand

SUMMARY:
UVA-1 has been reported to be beneficial to skin changes in scleroderma in several case reports and a few small studies. (Jacobe 2020) Interpretation of these reports has been difficult based on the small numbers of subjects involved and the non-blinded non-randomized nature of the reports. In a single controlled study with half-side comparison of 9 patients, the investigators could not demonstrate improvement with UVA-1 in the treated hand. (Thomas 2007) This study was limited by a small number of patients and the long disease duration prior to treatment (mean of 13 years). A more recent report of a patient with scleroderma for 2.5 years and severe acrosclerosis that responded to 21 sessions of UVA-1 with improved mobility and functionality renews interest in this treatment modality. (Cuenca-Barrales 2019)

In this trial patients will be randomized to have their dominant or non-dominant hand undergo 30 sessions of UVA1 therapy . We will assess patient's hand mobility, hand function, skin hardening (assessed by durometer measurements), skin thickness, as well as patient reported outcomes to determine efficacy.

This study will use a single-blind, prospective, randomized (dominant/non-dominant hand) comparator design to assess the effect of high dose (80-120 J/cm2) UVA1 therapy on hand function in scleroderma in a paired t-test design. This study will be placebo-controlled (with a UV-blocking gloved hand), cross-over, randomized clinical trial. Following the initial treatment period (30 treatments), patients will have the option to undergo the same high dose UVA1 treatment protocol on the untreated control hand. A follow up period of 12 months following completion of UVA1 therapy will prospectively follow patients to monitor for relapse of their disease to assess the durability of the clinical response to UVA1 therapy on hand scleroderma.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc), also called scleroderma, is a rare chronic autoimmune disease that can have a wide range of cutaneous, joint, and internal organ involvement. In the skin, SSc is characterized by enhanced fibroblast activity leading to hypertrophic dermal collagen that results in thickened, less flexible skin. (Hassani, 2016) SSc is often divided into two types based on extent of cutaneous involvement: diffuse SSc and limited SSc. The hand is a frequent area of involvement in both subtypes of SSc. Hand disability in SSc leads to a high burden on quality of life for patients as it limits both work and activities of daily living. Treatment for hand sclerosis remains limited with generally progressive disease despite aggressive treatment with anti-fibrotic medications, immunosuppressive agents, and topical approaches. Specific hand therapies include physiotherapy and injections of autologous adipose-derived stromal vascular fraction into the fingers with some success. (Guillaume-Jugnot, 2016; Liem, 2019)

Ultraviolet therapy has been used in dermatology for several decades. UVA-1 is a form of phototherapy that utilizes the longest wavelengths in the UV spectrum from 340-400 nm. It is able to penetrate deeper in the skin than other types of phototherapy and target different types of cells including fibroblasts. In sclerosing skin conditions UVA-1 appears to be superior to other forms of UV light. Medium to high dose UVA-1 also appears to be superior to low dose UVA-1 for sclerosing conditions. (Kreuter 2006).

UVA-1 has been reported to be beneficial to skin changes in SSc in several case reports and a few small studies. (Jacobe 2020) Interpretation of these reports has been difficult based on the small numbers of subjects involved and the non-blinded non-randomized nature of the reports. In a single controlled study with half-side comparison of 9 patients, the investigators could not demonstrate improvement with UVA-1 in the treated hand. (Thomas 2007) This study was limited by a small number of patients and the long disease duration prior to treatment (mean of 13 years). A more recent report of a patient with SSc for 2.5 years and severe acrosclerosis that responded to 21 sessions of UVA-1 with improved mobility and functionality renews interest in this treatment modality. (Cuenca-Barrales 2019)

If UVA1 therapy can significantly improve hand involvement in SSc with regards to functionality and disability, it may be a cost-effective and beneficial treatment for this patient segment with debilitating disease.

Purpose and Objectives:

1. To assess the efficacy of 30 sessions of ultraviolet-1 (UVA1) therapy in treating hand involvement of SSc in a prospective, randomized, investigator-blinded, intra-patient, UV-blocking glove-controlled, crossover clinical trial.

   1. To compare improvement in hand function as measured by the Hand Mobility in Scleroderma (HAMIS) test, in the UVA1-treated hand compared to control hand (gloved).
   2. To compare the improvement in hand function as measured by the Cochin hand functional disability scale (CHFDS) in the UVA1-treated hand compared to control hand (gloved).
   3. To compare the improvement in skin hardening based on durometer measurements in the UVA1-treated hand compared to control hand (gloved).
   4. To measure improvement in the physician measure of skin thickness on hands and fingers (0-3) scale after completion of 30 UVA1 sessions.
   5. To assess the duration of response after a complete 30-treatment course at 3 and12 months post treatment using the HAMIS, CHFDS, durometer, and physician skin thickness assessment.
2. Assess patient-reported outcomes before, during and after treatment using Skindex-16, Michigan Hand Questionnaire (MHQ), PROMIS-Physical Function (PROMIS-PF), Hand Disability in Systemic Sclerosis - Digital Ulcers(HDISS-DU) and Visual Analog Scale (VAS).

Study Design:

This study will use a single-blind, prospective, randomized (dominant/non-dominant hand) comparator design to assess the effect of high dose (80-120 J/cm2) UVA1 therapy on hand function in scleroderma in a paired t-test design. This study will be placebo-controlled (with a UV-blocking gloved hand), cross-over, randomized clinical trial. Following the initial treatment period (30 treatments), patients will have the option to undergo the same high dose UVA1 treatment protocol on the untreated control hand. A follow up period of 12 months following completion of UVA1 therapy will prospectively follow patients to monitor for relapse of their disease to assess the durability of the clinical response to UVA1 therapy on hand scleroderma.

Inclusion criteria:

* Must be able to understand and provide written informed consent
* Scleroderma skin involvement affecting both hands approximately equally
* Age of at least 18-years-old
* Male or female
* Ability to engage in twice weekly UVA1 sessions
* No changes in systemic therapy during the first 100 days of the study period

Exclusion criteria:

* On photosensitizing medication
* Inability to complete study visits
* UV light therapy in the 4 weeks prior to entering the study
* Commercial tanning or excessive sun exposure in the 4 weeks prior to entering the study
* Current pregnancy or planned pregnancy during the study period
* Use of topical therapies other than emollients (suprapotent corticosteroids) in the 2 weeks prior to entering the study
* History of intolerance to ultraviolet light
* Any other condition that will disqualify the patient from the study in the opinion of the investigator

Procedures:

This is a single-blinded, randomized, UV-blocking glove controlled, dominant/non-dominant hand, cross-over study to determine the efficacy of UVA1 in the treatment of hand scleroderma. Each participant will have at least one hand treated with UVA1 during the active treatment period of the study. The study will be performed at the University of Utah Dermatology Department using both the University of Utah E12 Clinic space as well as the Midvalley Clinic space. UVA1 lights boxes are located at both E12 and Midvalley locations. Personnel involved in the study will include the PI, the co-investigators, and the study coordinators. Approximately 27 patients will be enrolled to account for a 25% drop-out rate. The number needed to treat to show a difference in the treatment vs. control hands is 21. The study timeline is summarized in Table 1.

Screening:

For screening, subjects with qualifying scleroderma involving both hands will be asked to read and sign the informed consent document. They will be reminded that they are to take their time and, if necessary, take it home for further consideration. Questions will be answered. Those meeting inclusion / exclusion criteria who have signed informed consent will be enrolled.

After answering questions and prior to the first treatment the Principal Investigator (PI) will examine the entire patient and assess for the diagnosis of systemic sclerosis with bilateral hand involvement and perform the following assessments: HAMIS, CHFDS, durometer measurements, and mRSS. (Please see efficacy assessment section for details of HAMIS, CHFDS, durometer, and mRSS). Photographs of the hands and other affected areas will be taken. The patient will be asked to identify their dominant (writing) hand and their answer will be noted. Using a random number generator, the patient will be randomized to undergo UVA1 treatment vs UV-blocking glove (control) on the dominant hand. The non-dominant hand will receive the other modality. A study coordinator will perform the randomization on the day of first treatment and the PI will be blinded to the treatment assignment.

UVA1 Treatments:

Blinding:

A UV-blocking glove will be placed on the control hand as determined by the randomization process. Subjects will wear eyewear that occludes external light.

Evaluations for adverse effects will be carried out by the UVA1 operator (a nurse not involved in any assessments) and the blinded investigator at prescribed intervals. Evaluation of UVA1 efficacy on hand scleroderma will be assessed by a trained and experienced evaluator who is blinded as to the UVA1-treated side (covered / not covered). The efficacy evaluations will be carried out prior to treatments on days both evaluations and treatments are completed. After participants have been evaluated at the 3-month post-treatment study visit the blinded evaluator will become unblinded to the UVA1-treated side for the purpose of allowing participants to receive standard of care therapy. Therefore, participants will be allowed to receive additional UVA-1 treatments to one or both hands in addition to any other necessary standard of care treatments after the 3-month post-treatment visit.

Dosing Schedule:

Prior studies with UVA1 have shown that high and medium dose protocols (>40-120 J/cm2) are more effective than low dose (20-40 J/cm2) to treat sclerosing skin conditions. (Hassani, 2016) Thus, we will set the initiation dose at 50 J. The hands will be positioned approximately 9 inches from the bulbs. The palmar surface of the hand will be exposed for half the treatment and the dorsal surface for half the treatment. If tolerating well after three treatments, the dose will be increased to 60 J for three treatments and then 70 J for the remaining treatments.

Patients will return to clinic two-to-three times per week for 30 treatments over a 100-day period to receive UVA1 treatments. If the patient experiences redness, burning, pain, or blistering at the treatment site, treatment will be held if active symptoms persist at the time of the next scheduled treatment. If the symptoms have resolved and the patient has healed by the next scheduled treatment, the UVA1 energy will be reduced by 10 J of the previously delivered dose. Dose escalation will then proceed by increasing the UVA1 energy after three well tolerated treatments.

Evaluations:

1. Efficacy evaluations will be performed at baseline, after 15 UVA1 treatment sessions, after 30 UVA1 treatment sessions, and at 3 and 12 months after completion of all UVA1 treatments. For each evaluation prior to the 12-month evaluation, one of the sub-Investigators who is blinded to the treatment assignments will generate and record the HAMIS, CHFDS, Durometer, and mRSS. Hands will be photographed. Patients will complete all PROM including using Skindex-16, Michigan Hand Questionnaire (MHQ), PROMIS-Physical Function (PROMIS-PF), Hand Disability in Systemic Sclerosis - Digital Ulcers(HDISS-DU), and Visual Analog Scale (VAS).

The blinded evaluator will also perform safety evaluation and document study-related adverse events.

1. Primary Efficacy Measure:

   The efficacy will be measured using the HAMIS test score to assess for improvement over time and as compared to the untreated hand. The primary endpoint will be assessed after 30 UVA1 treatments. The primary endpoint is improvement in HAMIS score as compared to the untreated hand after 30 UVA1 treatment sessions.
2. Secondary Efficacy Measures:

Secondary efficacy measures include HAMIS test score improvement from baseline in treated and untreated hands after 30 UVA1 treatment sessions, as well as changes in CHFDS, Durometer measures, mRSS, Skindex-16, MHQ, PROMIS-PF, and VAS scores between baseline and after 30 UVA1 treatment sessions and (when applicable) between treated and untreated hands. Other secondary efficacy measures include change in HAMIS test scores CHFDS, Durometer measures, Physician assessment, Skindex-16, MHQ, PROMIS-PF, HDISS-DU, and VAS scores between completion of 30 UVA1 treatments and 3 and 12 months post-treatment in both hands as compared to baseline and after 30 UVA1 treatment sessions in each hand. Secondary endpoint measures also include time to disease worsening after treatment as defined by a 3-point (~10%) increase in HAMIS scores post-treatment.

Endpoint measure descriptions:

HAMIS is a hand function test developed for adults with systemic sclerosis. HAMIS consists of 9 items designed to measure all movements assessed in an ordinary range of motion (ROM)-measured hand test. Specific items test finger flexion and extension, thumb abduction, pincer grip, finger abduction/swelling, dorsal extension and volar extension of the wrist, and pronation and supination. Each item is graded on a 0-3 scale, where 0 corresponds to normal function and 3 denotes that the individual is unable to perform the item. Each hand is assessed separately. The minimum score for HAMIS is 0, representing normal hand function. The maximum score of HAMIS is 27, representing a high degree of dysfunction. (Sandqvist, 2000)

The CHFDS is a questionnaire with 18 questions concerning daily living activities, administered by a clinician, which each question scored on a scale from 0 (performed without difficulty) to 5 (impossible to do). The total score is obtained by adding the scores from all items (range 0-90), with lower scores indicating normal function and higher scores indicating poor function. This test was developed for rheumatoid arthritis but has been validated in scleroderma. (Rannaou, 2007)

A Durometer is an instrument for testing the hardness of various materials. It has been used in scleroderma to measure the hardness of affected skin as compared to normal skin.

The physician assessment on skin thickness on the hand and fingers based on the modified Rodnan skin score (mRSS) which is a standard outcome measure for skin disease in systemic sclerosis. The score is calculated by evaluating the skin thickness at 17 different body sites. Each site is graded from 0 to 3, with 0 representing normal skin and 3 representing severe skin thickness. The score is calculated by adding the scores at each site to arrive at a total score ranging from 0 (normal) to 51 (severe disease). (Khanna, 2017) In this study we will only calculate the score for the hands and fingers. Total possible score of 6 on each hand.

Skindex-16 is a 16-item validated assessment for the patient to identify the impact of their skin disease on three quality of life domains: symptoms, emotions, and physical functioning. Scores are normalized to a 0-100 scale with 0 representing no impact on quality of life and 100 representing maximal impact.

The Michigan Hand Questionnaire (MHQ) is a 37-item validated instrument exploring hand-specific outcomes across six domains: overall hand function, activities of daily living (ADLs), pain, work performance, aesthetics, and patient satisfaction with hand function. It asks questions separately about each hand, allowing for comparisons between hands. The raw score is converted to a 0-100 scale. For pain, a higher score indicates more pain, but for the other five scales, higher scores indicate better hand performance. The score for the affected hand is obtained by selecting either the right or the left hand score.

Hand Disability in Systemic Sclerosis - Digital Ulcers(HDISS-DU) is a patient reported outcome measure developed to capture the full spectrum of symptoms and disability related to digital ulcers, which are common and debilitating in scleroderma involving the hands. The instrument consists of 24 items. Responses are scored from 1 to 6 (6 scores), where 1 is 'yes, without difficulty', 2 is 'yes, with a little difficulty', 3 is 'yes, with some difficulty', 4 is 'yes with much difficulty', 5 is 'nearly impossible to do' and 'used unaffected hand only' (both responses were assigned the same score), and 6 is 'impossible'. The eighth response option 'did not do this activity in the past 7 days' is scored as missing. The overall HDISSDU score is calculated as the mean of non-missing item scores (with a missing data threshold of < 12 items) and ranged from a minimum score of 1 to a maximum score of 6, with increasing score corresponding to increasing disability.

PROMIS Physical Function (PROMIS-PF) is a computer adaptive test (CAT), wherein initial screening questions guide the need for additional questions following an iterative algorithm. For example, if a patient is unable to walk 100 feet without resting, an additional question about jogging 1 mile would not be asked. A weighted t-score results based on national averages with 50 as the mean score; >50 means higher physical function, <50 means lower physical function.

All PROs (Skindex-16, MHQ, PROMIS-PF) will be collected electronically at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand and provide written informed consent
* Scleroderma skin involvement affecting both hands approximately equally
* Age of at least 18-years-old
* Male or female
* Ability to engage in twice weekly UVA1 sessions
* No changes in systemic therapy during the first 100 days of the study period

Exclusion Criteria:

* On photosensitizing medication
* Inability to complete study visits
* UV light therapy in the 4 weeks prior to entering the study
* Commercial tanning or excessive sun exposure in the 4 weeks prior to entering the study
* Current pregnancy or planned pregnancy during the study period
* Use of topical therapies other than emollients (suprapotent corticosteroids) in the 2 weeks prior to entering the study
* History of intolerance to ultraviolet light
* Any other condition that will disqualify the patient from the study in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
HAMIS score of treated hand compared to the HAMIS score of the untreated hand after 30 UVA-1 treatments have been completed. | Approximately 100 days
  HAMIS graded on a 0-3 scale, where 0 corresponds to normal function and 3 denotes that the individual is unable to perform the item.

SECONDARY OUTCOMES:
Change in HAMIS score from baseline to after 30 UVA-1 treatments of treated hand. | Approximately 100 days
  HAMIS graded on a 0-3 scale, where 0 corresponds to normal function and 3 denotes that the individual is unable to perform the item.
Change in CHFDS score from baseline to after 30 UVA-1 treatments of treated hand. | Approximately 100 days
  The CHFDS is a questionnaire with 18 questions concerning daily living activities, administered by a clinician, which each question scored on a scale from 0 (performed without difficulty) to 5 (impossible to do). The total score is obtained by adding the scores from all items (range 0-90), with lower scores indicating normal function and higher scores indicating poor function. This test was developed for rheumatoid arthritis but has been validated in scleroderma. (Rannaou, 2007)
Change in skin hardness from baseline to after 30 UVA-1 treatments of treated hand. | Approximately 100 days
  A Durometer is an instrument for testing the hardness of various materials. It has been used in scleroderma to measure the hardness of affected skin as compared to normal skin.
Change in skin thickness from baseline to after 30 UVA-1 treatments of treated hand. | Approximately 100 days
  The physician assessment on skin thickness on the hand and fingers based on the modified Rodnan skin score (mRSS) which is a standard outcome measure for skin disease in systemic sclerosis. The score is calculated by evaluating the skin thickness at 17 different body sites. Each site is graded from 0 to 3, with 0 representing normal skin and 3 representing severe skin thickness. The score is calculated by adding the scores at each site to arrive at a total score ranging from 0 (normal) to 51 (severe disease). (Khanna, 2017) In this study we will only calculate the score for the hands and fingers. Total possible score of 6 on each hand.
Change in Skindex-16 score from baseline to after 30 UVA-1 treatments of treated hand. | Approximately 100 days
  Skindex-16 is a 16-item validated assessment for the patient to identify the impact of their skin disease on three quality of life domains: symptoms, emotions, and physical functioning. Scores are normalized to a 0-100 scale with 0 representing no impact on quality of life and 100 representing maximal impact.
Change in MHQ scores from baseline to after 30 UVA-1 treatments of treated hand. | Approximately 100 days
  The Michigan Hand Questionnaire (MHQ) is a 37-item validated instrument exploring hand-specific outcomes across six domains: overall hand function, activities of daily living (ADLs), pain, work performance, aesthetics, and patient satisfaction with hand function. It asks questions separately about each hand, allowing for comparisons between hands. The raw score is converted to a 0-100 scale. For pain, a higher score indicates more pain, but for the other five scales, higher scores indicate better hand performance. The score for the affected hand is obtained by selecting either the right or the left hand score.
Change in HDISS-DU from baseline to after 30 UVA-1 treatments of treated hand. | Approximately 100 days
  Hand Disability in Systemic Sclerosis - Digital Ulcers(HDISS-DU) is a patient reported outcome measure developed to capture the full spectrum of symptoms and disability related to digital ulcers, which are common and debilitating in scleroderma involving the hands. The instrument consists of 24 items. Responses are scored from 1 to 6 (6 scores), where 1 is 'yes, without difficulty', 2 is 'yes, with a little difficulty', 3 is 'yes, with some difficulty', 4 is 'yes with much difficulty', 5 is 'nearly impossible to do' and 'used unaffected hand only' (both responses were assigned the same score), and 6 is 'impossible'. The eighth response option 'did not do this activity in the past 7 days' is scored as missing. The overall HDISSDU score is calculated as the mean of non-missing item scores (with a missing data threshold of < 12 items) and ranged from a minimum score of 1 to a maximum score of 6, with increasing score corresponding to increasing disability.
Change in PROMIS-PF scores from baseline to after 30 UVA-1 treatments of treated hand. | Approximately 100 days
  PROMIS Physical Function (PROMIS-PF) is a computer adaptive test (CAT), wherein initial screening questions guide the need for additional questions following an iterative algorithm. For example, if a patient is unable to walk 100 feet without resting, an additional question about jogging 1 mile would not be asked. A weighted t-score results based on national averages with 50 as the mean score; >50 means higher physical function, <50 means lower physical function.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah MidValley Dermatology, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassani J, Feldman SR. Phototherapy in Scleroderma. Dermatol Ther (Heidelb). 2016 Dec;6(4):519-553. doi: 10.1007/s13555-016-0136-3. Epub 2016 Aug 12. PMID 27519050
- [Background] Sandler RD, Matucci-Cerinic M, Hughes M. Musculoskeletal hand involvement in systemic sclerosis. Semin Arthritis Rheum. 2020 Apr;50(2):329-334. doi: 10.1016/j.semarthrit.2019.11.003. Epub 2019 Nov 9. PMID 31812353
- [Background] Guillaume-Jugnot P, Daumas A, Magalon J, Jouve E, Nguyen PS, Truillet R, Mallet S, Casanova D, Giraudo L, Veran J, Dignat-George F, Sabatier F, Magalon G, Granel B. Autologous adipose-derived stromal vascular fraction in patients with systemic sclerosis: 12-month follow-up. Rheumatology (Oxford). 2016 Feb;55(2):301-6. doi: 10.1093/rheumatology/kev323. Epub 2015 Sep 8. PMID 26350489
- [Background] Liem SIE, Vliet Vlieland TPM, Schoones JW, de Vries-Bouwstra JK. The effect and safety of exercise therapy in patients with systemic sclerosis: a systematic review. Rheumatol Adv Pract. 2019 Dec 9;3(2):rkz044. doi: 10.1093/rap/rkz044. eCollection 2019. PMID 31858074
- [Background] Connolly KL, Griffith JL, McEvoy M, Lim HW. Ultraviolet A1 phototherapy beyond morphea: experience in 83 patients. Photodermatol Photoimmunol Photomed. 2015 Nov;31(6):289-95. doi: 10.1111/phpp.12185. Epub 2015 Jun 26. PMID 26052743
- [Background] Kroft EB, van de Kerkhof PC, Gerritsen MJ, de Jong EM. Period of remission after treatment with UVA-1 in sclerodermic skin diseases. J Eur Acad Dermatol Venereol. 2008 Jul;22(7):839-44. doi: 10.1111/j.1468-3083.2007.02576.x. Epub 2008 Apr 30. PMID 18452527
- [Background] Bongi SM, Del Rosso A, Galluccio F, Sigismondi F, Miniati I, Conforti ML, Nacci F, Cerinic MM. Efficacy of connective tissue massage and Mc Mennell joint manipulation in the rehabilitative treatment of the hands in systemic sclerosis. Clin Rheumatol. 2009 Oct;28(10):1167-73. doi: 10.1007/s10067-009-1216-x. Epub 2009 Jun 25. PMID 19554274
- [Background] Sandqvist G, Eklund M. Hand Mobility in Scleroderma (HAMIS) test: the reliability of a novel hand function test. Arthritis Care Res. 2000 Dec;13(6):369-74. PMID 14635312
- [Background] Khanna D, Furst DE, Clements PJ, Allanore Y, Baron M, Czirjak L, Distler O, Foeldvari I, Kuwana M, Matucci-Cerinic M, Mayes M, Medsger T Jr, Merkel PA, Pope JE, Seibold JR, Steen V, Stevens W, Denton CP. Standardization of the modified Rodnan skin score for use in clinical trials of systemic sclerosis. J Scleroderma Relat Disord. 2017 Jan-Apr;2(1):11-18. doi: 10.5301/jsrd.5000231. PMID 28516167
- [Background] Prasad S, Coias J, Chen HW, Jacobe H. Utilizing UVA-1 Phototherapy. Dermatol Clin. 2020 Jan;38(1):79-90. doi: 10.1016/j.det.2019.08.011. PMID 31753195
- [Background] Kreuter A, Hyun J, Stucker M, Sommer A, Altmeyer P, Gambichler T. A randomized controlled study of low-dose UVA1, medium-dose UVA1, and narrowband UVB phototherapy in the treatment of localized scleroderma. J Am Acad Dermatol. 2006 Mar;54(3):440-7. doi: 10.1016/j.jaad.2005.11.1063. Epub 2006 Jan 30. PMID 16488295
- [Background] Mouthon L, Poiraudeau S, Vernon M, Papadakis K, Perchenet L, Khanna D. Psychometric validation of the Hand Disability in Systemic Sclerosis-Digital Ulcers (HDISS-DU(R)) patient-reported outcome instrument. Arthritis Res Ther. 2020 Jan 6;22(1):3. doi: 10.1186/s13075-019-2087-4. PMID 31907061